CLINICAL TRIAL: NCT01123655
Title: Phase 1 Trial of CII APL A12 in Rheumatoid Arthritis Patients
Brief Title: Phase 1 Trial of Type II Collagen (CII) APL A12 in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMMA-007-08S
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): The study will have 3 treatment arms each with 10-12 patients who have demonstrated T cell immunity to CII and have an in vitro response to APL A12 at the screening visit. Patients will be randomized to one of the 2 treatment arms (30 micrograms APL A12 or placebo). Each of the 2 treatments will be given for 16 weeks.
  Intervention: Drug treatment will be stopped or interrupted if indicated and medical care will be given as appropriate.
  Intervention: Drug treatment will be stopped or interrupted if indicated and medical care will be given as appropriate.
  Interventions: Drug: APLA12; Drug: Placebo
- Arm 2 (Experimental): The next group will receive a higher dose (50 micrograms) and/or placebo (Block 2).
  Intervention: Drug treatment will be stopped or interrupted if indicated and medical care will be given as appropriate.
  Interventions: Drug: APLA12; Drug: Placebo
- Arm 3 (Experimental): Block 3 (Arm 3) will include placebo and both doses of APL/A12 to ensure 10-12 patients are enrolled in each arm ( total of approximately 32 subjects) so we will have 24 subjects who complete the 16 weeks of study treatment. Arms 2 and 3 will run simultaneously.
  Intervention: Drug treatment will be stopped or interrupted if indicated.
  Interventions: Drug: APLA12; Drug: Placebo

INTERVENTIONS:
Drug: APLA12 — Intervention: Drug treatment will be stopped or interrupted if indicated. Medical care will be provided at no cost to the patient.
Drug: Placebo — Drug treatment will be stopped or interrupted if indicated. Medical care will be provided at no cost to the patient.

SUMMARY:
This is a Phase I clinical trial to determine whether orally administered APL A12 at one or more doses is superior to placebo in effecting a 25% reduction in interferon (IFN) stimulation index in 1(II)-stimulated culture of peripheral blood mononuclear (PBMC) obtained from patients with Rheumatoid Arthritis (RA), which will be the primary outcome variable. In an effort to learn more about the mechanism of action of APL A12, the investigators will assess Th1/Th2/Th3 cytokine production in supernatants from 48h and 144h cultures of PBMC stimulated by 1(II) and by APL A12 above. The investigators will assess function of CD4+ CD25+ T regs to determine whether APL A12 improves their suppressive function. Flow cytometry combined with intracellular cytokine staining will be used in an effort to determine which T cell subset(s) is/are experiencing shifts in cytokine expression.

DETAILED DESCRIPTION:
The study will have 3 treatment arms each with 10 patients who have demonstrated T cell immunity to CII and have an in vitro response to APL A12 at the screening visit. Patients will be randomized to one of the 3 treatment arms. Each of the 3 treatments will be given for 16 weeks.

In keeping with a sequential dose escalation strategy, the originally proposed randomization scheme will be modified so that subjects will be randomized to receive either the lowest dose (30 mg) or placebo (Block 1), followed by the next dose (50 mg) or placebo (Block 2). We will begin with the lowest dose (30 g/day) and enroll 6 to receive 30 g/day APL A12 and 2 to receive placebo for 16 weeks. Results will be reported to the Data Monitoring Committee (DMC) for a decision to proceed to the next block based on indications of safety. If this dose does not cause adverse events or toxicity or worsens RA, we will proceed to enroll patients to receive 30 ug, or 50 g/day APL A12 or placebo for 16 weeks. A total of 32 subjects will be randomized to obtain 24 subjects who complete the study. Recruitment was difficult. Only 22 patients were randomized. There were not enough 50mcg patients enrolled so 2 treatment groups was analyzed. Arm 1 included 30 and 50 mcg and Arm 2 represents the patients that received placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for participation in the study.

* Male or female; age > 18 years.
* American College of Rheumatology (ACR) 1988 revised criteria for rheumatoid arthritis.
* Onset of disease age 16 or older.
* Onset of disease at least 3 months prior to enrollment.
* RA patients ages 18-85 with RA of 3 month duration which in the opinion of the examining rheumatologist is "clinically stable" and will likely not require adjustment of doses of Disease-modifying antirheumatic drugs (DMARDS), NSAIDS, prednisone, anti-tumor necrosis factor (anti-TNF) alpha therapies for the 16 weeks of the treatment phase of the study.
* Patients must agree to discontinue all "herbal remedies" as described in this protocol.
* Women of childbearing age will be advised to use effective means of contraception for the treatment phase of the trial and for 90 days thereafter. They must have a negative urine pregnancy test at the randomization visit. (Required by the FDA.)
* Men will be advised to use effective means of contraception for the treatment phase of the trial and for 90 days thereafter. (Required by the FDA.)
* Crohn's Disease Activity Index (CDAI) less than or equal to 30 at the baseline visit.
* Patients with a past history of malignant neoplasm will be eligible if they are 1 or greater years with no recurrence of malignant neoplasm.

Exclusion Criteria:

* Inability to render an informed consent in accordance with institutional guidelines.
* Participation in another clinical research study involving the evaluation of another investigational drug within 90 days of entry into this study.
* RA patients on >7.5 mg prednisone a day.
* RA patients with intra-articular corticosteroid injections during the previous 30 days.
* Concurrent serious medical condition which in the opinion of the investigator makes the patient inappropriate for the study. Hepatitis B abd/or C patients with inactive disease (as determined by PI) will be enrolled.
* Positive urine pregnancy test
* Age 85 years or greater.
* Use of "fish oil" within the previous 4 weeks of the baseline visit.
* Therapy consisting of auranofin or cyclophosphamide (all other DMARDs are allowed).
* Previous autologous or heterologous stem cell transplantation.
* Active malignant neoplasm or past treatment for malignant neoplasm 1 year from screening visit.
* Use of oral CII within the past 1 year. (Since oral tolerance is short-lived, we will permit patients in the study who have been off oral CII for > 1 year)
* Diabetes requiring insulin or on oral medications must be well managed at baseline. Adjustment of insulin or on oral medications will be allowed during the study.
* Serum creatinine 2.0 mcg/dL.
* An 1(II) IFN value <100% of the PBS IFN value within 1 month or less prior to the baseline and less than 25% reduction in APL A12 + 1(II) IFN from 1(II) IFN concentration.
* CDAI > 30 at the baseline visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold E Postlethwaite, MD, Principal Investigator — Memphis VA Medical Center, Memphis, TN
Locations (1):
- Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 1, 2009-September 30, 2015.
Groups:
- 30 mcg of APL/Day: 30 micrograms compared with placebo
- 50 ug APL/Day: 50 mcg and 30mcg compared to placebo
- Placebo: Placebo group
Period: Overall Study
Arm/Group | 30 mcg of APL/Day | 50 ug APL/Day | Placebo
Started | 10 | 4 | 8
Completed | 9 | 3 | 7
Not Completed | 1 | 1 | 1
Not completed — Medication for RA had to be changed | 1 | 0 | 0
Not completed — new illness | 0 | 1 | 0
Not completed — began prohibitive drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients with rheumatoid arthritis who had an immunity demonstrated to type II collagen who were unable to be reduced in in vitro culture by APL A12.
  30 and 50 mcg/day doses were combined because animal data showed no difference between doses.
Groups:
- 30 or 50 ug APL/Day: The study will have 3 treatment arms each with 10-12 patients who have demonstrated T cell immunity to CII and have an in vitro response to APL A12 at the screening visit. Patients will be randomized to one of the 3 treatment arms. Each of the 3 treatments will be given for 16 weeks.
  In keeping with a sequential dose escalation strategy, the originally proposed randomization scheme will be modified so that subjects will be randomized to receive:
  either the lowest dose (30 micrograms) or placebo (Block 1). We will begin with the lowest dose (30 micrograms/day) and enroll 6 to receive 30 micrograms/day APL A12 and 2 to receive placebo for 16 weeks. Results will be reported to the DMC for a decision to proceed to the next block based on indications of safety APL A12: IND 103860: The study drug APL A12 is a man made (or synthesized) fragment similar to a portion of natural type II collagen, the major collagen found in joint cartilage. Cartilage is the tough, elastic tissue found in
- Placebo: Block 3 (Arm 3) will include placebo and both doses of APL/A12 to ensure 10-12 patients are enrolled in each arm ( total of approximately 32 subjects) so we will have 24 subjects who complete the 16 weeks of study treatment. Arms 2 and 3 will run simultaneously.
  APL A12: IND 103860: The study drug APL A12 is a man made (or synthesized) fragment similar to a portion of natural type II collagen, the major collagen found in joint cartilage. Cartilage is the tough, elastic tissue found in various parts of the body, including the joints. The best dose of APL A12 to use in patients with rheumatoid arthritis is not known.
- Total: Total of all reporting groups
Arm/Group | 30 or 50 ug APL/Day | Placebo | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.08 (8.47) | 65.8 (9.91) | 63.94 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All southern region residents
  Participants
    United States | 14 | 8 | 22
Immunity to Type-II collagen and in vitro decrease by APL12 [Count of Participants; unit: Participants] — We could not analyze all the patients due to adverse events, drop outs or not all participants had data available for all measurements.
  Participants | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number and Percent of Participants With Reduction of Immunity to Collagen Type-II After APLA-12 Treatment.
Description: The primary outcome variable is the presence of a > 25% reduction in net IFN concentration in supernatants of 1(II)-stimulated PBMC cultures from baseline after 16 weeks of treatment.
Time Frame: 16 weeks
Population: We could not analyze all the patients due to adverse events, drop outs or not all participants had data available for all measurements
Measure: Count of Participants; unit: Participants
Groups:
- APL 30 and 50ug/Day: 30ug and 50ug/ day were combined for analysis and were combined because the period of funding expired before all the proposed number of patients could be enrolled for the 50ug/day Arm.
  APL A12: IND 103860: The study drug APL A12 is a man made (or synthesized) fragment similar to a portion of natural type II collagen, the major collagen found in joint cartilage. Cartilage is the tough, elastic tissue found in various parts of the body including the joints. The best dose of APL A12 to use in patients with RA is not known.
- Placebo: Block 3 (Arm 3) will include placebo.
  Dose of placebo was 2ml of IV saline.
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 10 | 6
Participants | 9 | 4
Statistical Analysis 1: Comparison: APL 30 and 50ug/Day vs Placebo; Specified to be a reduction from baseline values of net IFNƔ concentration of ≥ 25% in αl(ll)-stimulated PBMC culture supernatants (calculated as αI(II)-IFNƔ-PBS IFNƔ in patients receiving APL A12 compared to placebo; Test type: Equivalence — P less than 0.05 was the criteria for equivalence; p = 0.5179, Fisher Exact
Statistical Analysis 2: Comparison: APL 30 and 50ug/Day; Test type: Equivalence — Null hypothesis was that the response rate in the APL treated groups is not significantly difference from the 50% spontaneous response rate; p = 0.0114, Exact Test
Statistical Analysis 3: Comparison: Placebo; Test type: Equivalence — Null hypothesis was that the response rate in the placebo group is not significantly difference from the 50% spontaneous response rate; p = 0.4142, Exact Test

2. Secondary Outcome: Flow Cytometry
Description: Change in Percentage of CD4+CD25+FoxP3 T regulatory cells, CD4+IL-10+ cells, CD4+ IL-4+ cells, CD4+IL17+ cells. Some patients had only had enough blood collected at 8 weeks or 16 weeks or dropped out after 8 weeks, and we used/combined what was available.
Time Frame: baseline and 8 or 16 weeks
Population: Not all participants had data available for all measurements.
Measure: Mean (Standard Deviation); unit: percent change in number of cells
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent change in number of cells
  CD4+IL-4+: number analyzed (Participants) | 9 | 3
  CD4+IL-4+ | 0.8959 (1.0736) | 1.9400 (2.8626)
  CD4+CD25hi+FoxP3: number analyzed (Participants) | 10 | 4
  CD4+CD25hi+FoxP3 | 3.4240 (4.3569) | 0.9600 (3.4390)
  CD4+IL-17+: number analyzed (Participants) | 10 | 3
  CD4+IL-17+ | 1.5299 (4.1486) | -0.4230 (2.1367)
  CD4+IL-10+: number analyzed (Participants) | 10 | 4
  CD4+IL-10+ | 0.1735 (0.5400) | 0.3385 (0.4444)

3. Secondary Outcome: Clinical Disease Activity Index (CDAI) at 0 and 16 Weeks Follow up
Description: Interpretation of Clinical Disease Activity Index (CDAI) scores < 2.8 indicate remission; >2.8 and <= 10 indicates low disease activity; >10 and <= 22 indicates moderate disease activity; >22 indicates high disease activity.
Time Frame: 0 and16 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: disease activity score
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 14 | 8
disease activity score
  CDAI at 0 weeks | 10.0333 [0.7 to 12.5] | 10.3271 [2.4 to 23]
  CDAI at 16 weeks: number analyzed (Participants) | 10 | 4
  CDAI at 16 weeks | 9.8778 [1.1 to 29.5] | 12.8000 [6.7 to 19.5]
Statistical Analysis 1: Comparison: APL 30 and 50ug/Day vs Placebo; Test type: Equivalence — P greater than 0.05 was the criteria for equivalence; p > 0.05, Mixed Models Analysis — P value is applicable for baseline and follow-up data

4. Secondary Outcome: Change in Cytokine Profile From Baseline and 16 Weeks
Description: Cytokines assessed are IL-10, IL-13, IL-5, IL-1B, IL-9, IL-17A, IL-6, IL-21, TGF-B, TNFa,and MIP3A.
Time Frame: 0 and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: absolute change (picograms/milliliter)
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
absolute change (picograms/milliliter)
  IL-10 | -22.51 (82.57) | -4.70 (5.99)
  IL-13 | -6.46 (17.12) | -0.83 (4.57)
  IL-5 | 5.19 (19.11) | -2.42 (2.34)
  IL-1B | 617.1 (2111.8) | 45.64 (280.1)
  IL-9 | 196.1 (679.2) | -45.37 (56.10)
  TGF-B1 | 0.12 (0.42) | -0.06 (0.41)
  IL-17A | -104.2 (229.9) | 5.4091 (7.4381)
  IL-6 | -2002.9 (10752.9) | 3.97 (261.4)
  TNFa | -7.50 (39.98) | 0.30 (4.14)
  IL-21 | -4.32 (10.92) | 218.3 (492.9)
  MIP3A(CCL-20) | -36.39 (89.60) | 3.60 (21.08)
Statistical Analysis 1: Comparison: APL 30 and 50ug/Day vs Placebo; Test type: Equivalence — p value greater than 0.05 was the criteria for equivalence; p > 0.05, t-test, 2 sided — P value is applicable to IL-17a, IL-10, IL-1b, IL-9, IL-13, IL-5, IL-21, IL-6, TNFa, TGFb, MIP3a

5. Secondary Outcome: Change in IgG and IgA Immunoglobulin From Baseline to 8 or 16 Weeks
Description: The change was computed between baseline and 8 or 16 weeks, whichever was available.
Time Frame: baseline and 8 or 16 wks
Population: Some participants only had measurable data at 8 weeks, or dropped out before 16 weeks.
Measure: Mean (Standard Deviation); unit: absolute change (followup-baseline) ng/m
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 10 | 4
absolute change (followup-baseline) ng/m
  change in IgG | 1047.01 (3570.28) | 11.43 (109.27)
  change in IgA | 3410.3 (11339.8) | 103.69 (233.92)

6. Secondary Outcome: Neutrophils Counts at 0 and 16 Weeks
Description: Laboratory Results of A12 vs Placebo:Complete blood count Neutrophil count to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent of total number of blood cells
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent of total number of blood cells
  0 weeks Neutrophils | 60.9 (2.4) | 60 (3.2)
  16 weeks Neutrophils | 59.2 (2.6) | 62.4 (3.5)

7. Secondary Outcome: A12 Treated vs Placebo of Monocytes.
Description: Laboratory Results of A12 treated vs Placebo of Monocytes to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: Baseline and 16 wks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent of total white blood cells
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent of total white blood cells
  Baseline | 9.1 (0.7) | 9.25 (0.9)
  16 weeks | 8.93 (0.7) | 7.53 (1)

8. Secondary Outcome: Eosinophils
Description: Laboratory Results of A12 treated vs Placebo of Eosinophils to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent in total white blood cells
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent in total white blood cells
  Baseline | 2.29 (0.5) | 4.4 (0.7)
  16 weeks | 2.69 (0.6) | 4.11 (0.7)

9. Secondary Outcome: Laboratory Results of A12 vs Placebo: Lymphocytes
Description: Measure to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent in total white blood cells/ml
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent in total white blood cells/ml
  0 Week Lymphocytes | 26.92 (2.22) | 25.41 (2.94)
  16 weeks Lymphocytes | 28.2 (2.35) | 25.37 (3.1)

10. Secondary Outcome: Laboratory Results of A12 vs Placebo: Basophils
Description: as for outcome 9
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent in total white blood cells/ml
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent in total white blood cells/ml
  0 week-Basophils | 0.53 (0.09) | 0.6 (0.12)
  16 week Basophils | 0.67 (0.097) | 0.47 (0.13)

11. Secondary Outcome: Hematocrit
Description: Laboratory Results of A12 vs Placebo to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio of RBC to total blood cells/volume
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
ratio of RBC to total blood cells/volume
  0 week HCT | 40.63 (0.85) | 42 (1.13)
  16 week HCT | 39.69 (0.9) | 42.6 (1.19)

12. Secondary Outcome: Laboratory Results of A12 vs Placebo-Total Immunoglobulin (Immature Granulocytes)
Description: as for outcome 9
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams per deciliter
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
grams per deciliter
  0 week-IG | 0.3 (0.05) | 0.24 (0.06)
  16 week-IG | 0.3 (0.05) | 0.33 (0.07)

13. Secondary Outcome: Red Blood Cell Distribution Width (RDW)
Description: Laboratory Results of A12 vs Placebo RDW is a measure of the range of variation of red blood cell volume reported as part of a standard blood count to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: 0 and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent of mean corpuscular volume
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
percent of mean corpuscular volume
  Baseline-RDW | 14.67 (0.31) | 14.15 (0.41)
  16 week RDW | 14.8 (0.33) | 13.9 (0.43)

14. Secondary Outcome: Hemaglobin
Description: as for outcome 11
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams/deciliter
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
grams/deciliter
  Baseline -Hgb | 13.66 (0.29) | 14.23 (0.38)
  16 week Hgb | 13.31 (0.3) | 14.31 (0.4)

15. Secondary Outcome: Red Blood Cells
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: 10^6 cells/uL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
10^6 cells/uL
  0 week RBC | 4.66 (0.13) | 4.49 (0.17)
  16 week RBC | 4.6 (0.13) | 4.57 (0.17)

16. Secondary Outcome: White Blood Count
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: 10^3 cells/uL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
10^3 cells/uL
  0 week WBC | 7.24 (0.43) | 5.88 (0.57)
  16 week WBC | 7.26 (0.47) | 6.23 (0.61)

17. Secondary Outcome: Platelets
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: 10^3 cells/uL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
10^3 cells/uL
  0 week Platelet | 248.71 (14.81) | 224.5 (19.6)
  16 week Platelet | 256.96 (15.51) | 225.44 (20.43)

18. Secondary Outcome: AST, ALT and Alkaline Phosphatase
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
IU/L
  0 week-AST | 32.29 (3.36) | 39.75 (3.97)
  16 week AST | 31.61 (3.67) | 33.52 (4.52)
  0 week ALT | 28.8 (3.2) | 35.75 (3.94)
  16 week ALT | 26.21 (3.33) | 35.62 (4.24)
  0 week alkaline phos | 97.79 (5.05) | 70.75 (6.13)
  16 week alkaline phos | 86.64 (5.34) | 73.07 (6.72)

19. Secondary Outcome: Ca, BUN, Glucose,Creatinine, Total Bilirubin
Description: Laboratory Results of A12 vs Placebo-CMP to determine whether APL has any effect on routine blood counts, chemistries, electrolytes, immunoglobulin to measure potential toxicities
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
mg/dl
  0 week calcium | 9.35 (0.09) | 9.11 (0.11)
  16 week calcium | 9.2 (0.1) | 9.22 (0.12)
  0 week BUN | 15.7 (2.37) | 15.37 (2.93)
  16 week BUN | 17.32 (2.45) | 15.56 (3.13)
  0 week glucose | 109.4 (9.71) | 112.4 (11.9)
  16 week glucose | 92.67 (10.2) | 86.72 (12.9)
  0 week total bilirubin | 0.68 (0.067) | 0.63 (0.082)
  16 week total bilirubin | 0.53 (0.7) | 0.75 (0.088)
  0 week creatinine | 0.945 (0.208) | 0.811 (0.244)
  16 week creatinine | 1.0050 (22.96) | 0.8501 (0.2818)

20. Secondary Outcome: Sodium, Potassium and Chloride
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
mmol/L
  0 week sodium | 140.7 (0.8) | 140.25 (0.98)
  16 week sodium | 141.46 (0.84) | 140.34 (1.06)
  0 week potassium | 3.9 (0.16) | 4 (0.2)
  16 week potassium | 3.8 (0.17) | 4.03 (0.2)
  0 week chloride | 102.9 (0.73) | 100.75 (0.88)
  16 week chloride | 103.22 (0.78) | 100.9 (0.97)

21. Secondary Outcome: Total Protein, Albumin
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
g/dL
  0 week total protein | 7.75 (0.17) | 7.64 (0.2)
  16 week total protein | 7.16 (0.19) | 7.8 (0.2)
  0 week albumin | 4.18 (0.08) | 4.22 (0.098)
  16 week albumin | 4.16 (0.084) | 4.42 (0.11)

22. Secondary Outcome: C-reactive Protein
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
mg/L
  0 week CRP | 11.8 (3.13) | 10.57 (4.61)
  16 week CRP | 11.38 (3.07) | 8 (4.61)

23. Secondary Outcome: Rheumatoid Factor
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
IU/mL
  0 week RF | 36.72 (9.4) | 23.75 (14.15)
  16 week RF | 25.29 (9.4) | 23.35 (14.15)

24. Secondary Outcome: Sedimentation Rate
Description: as for outcome 11
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm/hr
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
mm/hr
  0 week ESR | 30.85 (5.13) | 18.62 (6.7)
  16 week ESR | 33.5 (5.29) | 20.26 (6.9)

25. Secondary Outcome: Laboratory Results of A12 vs Placebo Anti-CCP Antibody
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
IU/mL
  0 week anti CCP | 310.6 (35.2) | 127.54 (44.9)
  16 week anti CCP | 319.07 (35.63) | 120.9 (45.52)

26. Secondary Outcome: Patient Global Assessment (PGA) and Physician Global Assessment
Description: Patient and Physician (PI) Assessments both range from 0-10 with 10 being the most disease activity
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
score on a scale
  0 week PI Assessment | 2.6 (0.46) | 3.26 (0.77)
  16 week PI Assessment | 2.77 (0.5) | 4.3 (0.7)
  0 week Patient Assessment | 3.99 (0.52) | 4.8 (0.9)
  16 week Patient Assessment | 4.7 (0.59) | 3.75 (0.78)

27. Secondary Outcome: Modified Health Assessment Questionnaire (MHAQ)
Description: Modified Health Assessment Questionnaire (MHAQ) 0-8 with 8 being the most activity
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: MHAQ units on a scale
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
MHAQ units on a scale
  0 week MHAQ | 3.44 (1.14) | 1.75 (1.71)
  16 week MHAQ | 4 (1.14) | 2.5 (1.9)

28. Secondary Outcome: Duration of Morning Stiffness in Joints
Description: Duration of morning stiffness in the joints, in minutes.
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
minutes
  0 week stiffness | 64.49 (98.81) | 38.75 (140.22)
  16 week stiffness | 184.44 (93.48) | 54.78 (195.3)

29. Secondary Outcome: CDAI
Description: Clinical Disease Activity Index (CDAI) 0-76 mm. Interpretation of CDAI scores < 2.8 indicate remission; >2.8 and <= 10 indicates low disease activity; >10 and <= 22 indicates moderate disease activity; >22 indicates high disease activity.
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
centimeters
  0 week CDAI | 10 (2) | 10.3 (3.3)
  16 week CDAI | 9.9 (2.2) | 12.8 (3)

30. Secondary Outcome: Vital Signs-Temperature
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: degrees Fahrenheit
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
degrees Fahrenheit
  0 week temperature | 97.4 (0.19) | 98 (0.25)
  16 week temperature | 97.4 (0.2) | 97.83 (0.27)

31. Secondary Outcome: Vital Sign - Pulse
Description: heartbeats per minute
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
beats per minute
  0 week pulse | 73.8 (3.23) | 72.46 (4.34)
  16 week pulse | 74.74 (3.47) | 71.83 (4.6)

32. Secondary Outcome: Weight
Description: Weight in kg
Time Frame: 0-16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
kilograms
  0 week weight | 84.06 (3.17) | 93.5 (4)
  16 week weight | 83 (3.18) | 95.21 (4)

33. Secondary Outcome: Vitals - Blood Pressure
Description: measurement of blood pressure (mmHg)
Time Frame: 0 weeks and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
mm Hg
  0 week BP systolic | 134.85 (3.9) | 131.51 (5.2)
  16 week BP systolic | 130.35 (4.2) | 140.67 (5.5)
  0 week diastolic | 77.23 (2.53) | 71.13 (3.4)
  16 week diastolic | 76.9 (2.74) | 74.75 (3.67)

34. Secondary Outcome: Vitals - Respirations
Description: Respirations represents breaths per minute
Time Frame: 0 weeks and 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | APL 30 and 50ug/Day | Placebo
Number analyzed (Participants) | 12 | 5
breaths per minute
  0 weeks | 18.3 (0.63) | 18.84 (0.5)
  16 weeks | 18.54 (0.4) | 17.7 (0.5)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- 30 ug and 50 ug APL/Day: 30 micrograms APL A12/day and 50 micrograms APL A12/day
  APL A12: IND 103860: The study drug APL A12 is a man made (or synthesized) fragment similar to a portion of natural type II collagen, the major collagen found in joint cartilage. Cartilage is the tough, elastic tissue found in various parts of the body, including the joints. The best dose of APL A12 to use in patients with rheumatoid arthritis is not known.
- Placebo: Block 3 (Arm 3) will include placebo
  Dose was 2ml of IV saline.
Arm/Group | 30 ug and 50 ug APL/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/8
Other Adverse Events (participants affected / at risk) | 8/14 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 ug and 50 ug APL/Day (N=14) | Placebo (N=8)
cardiac arrest (Cardiac disorders) | 1 (1) | 0
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — hospitalized
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 ug and 50 ug APL/Day (N=14) | Placebo (N=8)
malaise, itching (Immune system disorders) | 1 (1) | 0 (0)
flu-GI virus (Immune system disorders) | 2 (2) | 0 (0)
RA flare (Immune system disorders) | 1 (1) | 0 (0)
Burning rash on cheek (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
lips tingling (Nervous system disorders) | 0 (0) | 1 (1)
lightheaded with ringing in ears (General disorders) | 0 (0) | 1 (1)
injection site infection (Infections and infestations) | 1 (1) | 0 (0)
sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pet bite (Infections and infestations) | 1 (1) | 0 (0)
l4-l5 decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
broken tooth (General disorders) | 1 (1) | 0 (0)
lesion removed from ear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
sinusitis (General disorders) | 0 (0) | 1 (1)
atypical chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sore throat (General disorders) | 0 (0) | 1 (1)
bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lipoma removal (Surgical and medical procedures) | 0 (0) | 0 (0)
DJD worse (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes